CLINICAL TRIAL: NCT01609920
Title: Non-invasive Nodal Staging in Breast Cancer With Magnetic Resonance Imaging Lymphography Using Gadofosveset
Brief Title: Nodal Staging in Breast Cancer With MRL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer recently halted production of gadofosveset.
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-2-032
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2013-05

CONDITIONS: Breast Neoplasms
Keywords: MRI; lymph node metastases; breast cancer; gadofosveset
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis | interventions — gadofosveset trisodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadofosveset MRL (Experimental)
  Interventions: Drug: Gadofosveset enhanced MRL of axillary lymph nodes

INTERVENTIONS:
Drug: Gadofosveset enhanced MRL of axillary lymph nodes — A MRL of the axilla will be performed before and after administration of a single IV bolus injection of gadofosveset of an equivalent of 0.03 mmol Gd/kg body weight at an injection speed of 1.5 mL/sec., followed by a saline flush of 25 mL at an injection speed of 1.5 mL/sec.
  Other Names: Vasovist; Ablavar; Gadofosveset

SUMMARY:
The aim of this study is to examine the diagnostic performance of gadofosveset enhanced magnetic resonance imaging lymphography (MRL).

The diagnostic performance of MRL will be determined on the basis of a node-to-node matching of imaged nodes to the definitive histopathology. The pathologic examination of the sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND) will be regarded as the golden standard for nodal involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient with histopathologically confirmed breast cancer about to undergo nodal staging.
2. Willing and able to undergo all study procedures
3. Has personally provided written informed consent.

Exclusion Criteria:

1. Age <18,
2. Pregnancy
3. Contra indications for MRL such as pacemaker, aneurysm clips or severe claustrophobia.
4. Allergy to any of the ingredients of Gadofosveset (Vasovist® /Ablavar®)
5. Being unable to give informed consent in person
6. Acute or chronic severe renal insufficiency (glomerular filtration rate <45 mL/min/1.73m2)1.
7. Acute renal insufficiency of any severity due to the hepato-renal syndrome.
8. Known (or suspicion of) QT- prolongation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The diagnostic performance (sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV)) of axillary MRL in predicting the involvement of metastases | Participants will be followed from the moment of first out-hospital clinic vistit untill final breast surgery, an expected average of 4 weeks.
  The main study parameter will be the diagnostic performace (sensitivity, specificity, NPV and PPV) of the axillary MRL in predicting the involvement of metastases in the investigated lymph nodes. Each node will be scored on MRL as 0= benign, 1=malign. These results will be compared with the histopathological results of the SNLB procedure of ALND procedure on an node by node basis. So the diagnostic performace can be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: R.G.H. Beets-Tan, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center (MUMC) AZM, Maastricht, Limburg, Netherlands